CLINICAL TRIAL: NCT01054521
Title: A Randomized Comparison Study of Temperature-controlled and Bipolar Radiofrequency for Inferior Turbinate Reduction in Patients With Chronic Rhinitis
Brief Title: A Randomized Study of Temperature-controlled and Bipolar Radiofrequency for Inferior Turbinate Reduction
Acronym: CompareRFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: wbanhiran
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Patients With Chronic Rhinitis Who Failed Medical Treatment
Keywords: radiofrequency turbinate reduction; nasal obstruction; Temperature-controlled radiofrequency; Bipolar radiofrequency; chronic rhinitis.
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temperature-controlled RF (TCRF) (Experimental): The temperature-controlled RF was done under local anesthesia (0.5% xylocaine with adrenaline 1:200,000 injection at both inferior turbinates.) The RF probe will be inserted at inferior turbinate for 5 points both left and right nasal cavity (2 at anterior end, 2 at middle part and 1 at posterior end). We apply energy of 300 J, 85 C, and 15 W each point. After procedures the patients was observed at 1 hour before discharge without any packings.
  Interventions: Procedure: Temperature-controlled RF
- Bipolar RF (BRF) (Active Comparator): The bipolar RF (BRF) probe will be inserted at the same area with TCRF. We use 2.5 watt and 3 sec for each point but will stop immediately if the burning color or sound are detected. Otherwise was the same with TCRF.
  Interventions: Device: Bipolar RF

INTERVENTIONS:
Procedure: Temperature-controlled RF — The temperature-controlled RF was done under local anesthesia (0.5% xylocaine with adrenaline 1:200,000 injection at both inferior turbinates.) The RF probe will be inserted at inferior turbinate for 5 points both left and right nasal cavity (2 at anterior end, 2 at middle part and 1 at posterior end). We apply energy of 300 J, 85 C, and 15 W each point. After procedures the patients was observed at 1 hour before discharge without any packings.
  For nontemperature-controlled RF, the probe will be inserted at the same area with TCRF. We use 2.5 watt and 3 sec for each point but will stop immediately if the burning color or sound are detected. Otherwise was the same with TCRF.
  Other Names: Temperature-controlled RF device is Gyrus ENT.
  Arms: Temperature-controlled RF (TCRF)
Device: Bipolar RF — The bipolar RF probe will be inserted at the same area with TCRF. The energy used will be 2.5 watt and 3 sec for each point but will stop immediately if the burning color or sound are detected. Otherwise was the same with TCRF.
  Other Names: Bipolar RF device is Select Sutter.
  Arms: Bipolar RF (BRF)

SUMMARY:
Currently, there are several alternative treatments for patients with chronic rhinitis (CR) who failed medication. Although, most of the researches have been focusing on temperature-controlled RF (TCRF), the cost is a major limitation for applying it worldwide. The investigators objective of this study is to compare the subjective and objective outcomes of Bipolar RF (BRF) with the more popular TCRF for CR treatment. The investigators hypothesized that both have equivalent outcomes but with less operative time and potentially at lower cost.

ELIGIBILITY:
Inclusion Criteria:

* Adults with snoring and chronic nasal obstruction.
* Respond to topical decongestant but not respond to nasal steroids, oral anti-histamine and oral decongestant
* Consent to the protocol.

Exclusion Criteria:

* Chronic active sinusitis, severe Deviated nasal septum (DNS), nasal polyps, sinonasal tumor, previous sinonasal surgery or head neck irradiation.
* Uncontrolled bleeding disorders, hypertension, or cardiovascular diseases
* Not complete the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog scale scores of nasal obstructive symptom. | Up to 1 year follow-up

SECONDARY OUTCOMES:
VAS scores of nasal discharge, sneezing, hyposmia, postnasal drip | Up to 1 year follow-up
  Shor-term at 4th week and long-term at 1 year follow-up
Postoperative crust, mucociliary transportation time (MTT), minimal cross sectional area (MCA), total nasal volume (VOL), nasal airway resistance (NAR) at 75 Pa | Up to 1 year follow-up
  Crusting was assessed at 1st week and 4th week, MTT at 4th week, and MCA, VOL, and NAR were assessed before and after treatment at 4th week and one year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wish Banhiran, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Banhiran W, Assanasen P, Tantilipikorn P, Nujchanart N, Voraprayoon S, Bunnag C. A randomized study of temperature-controlled versus bipolar radiofrequency for inferior turbinate reduction. Eur Arch Otorhinolaryngol. 2015 Oct;272(10):2877-84. doi: 10.1007/s00405-014-3410-y. Epub 2014 Nov 29. PMID 25432641